CLINICAL TRIAL: NCT01371149
Title: A Clinical Trial to Optimise Patient-ventilator Interaction in Patients With Chronic Respiratory Failure
Brief Title: Patient -Ventilator Interaction in Chronic Respiratory Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michelle Ramsay (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, Michelle Ramsay, Dr, Guy's and St Thomas' NHS Foundation Trust
Organization: Guy's and St Thomas' NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10/H0716/67
Record Dates: First submitted 2011-06-09; First posted 2011-06-10 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Hypercapnic Respiratory Failure; Obesity Hypoventilation Syndrome; Neuromuscular Disease; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Obesity Hypoventilation Syndrome; Neuromuscular Diseases; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physician led ventilator set up (No Intervention): Patients will be set up on non-invasive ventilation as per the current gold standard physician led approach
- parasternal electromyography (EMG) set up (Experimental): Ventilation parameters will be manipulated and titrated according to physiological measurements including signal from parasternal EMG and patient- ventilator asynchrony.
  Interventions: Other: Surface parasternal electromyography (EMG) set up

INTERVENTIONS:
Other: Surface parasternal electromyography (EMG) set up — Ventilation parameters will be manipulated and titrated according to physiological measurements including signal from parasternal EMG and patient- ventilator asynchrony.
  Arms: parasternal electromyography (EMG) set up

SUMMARY:
To evaluate a novel advanced physiological monitoring system to improve nocturnal non-invasive ventilation (NIV) in Neuromuscular disease (NMD), Chest wall disease (CWD), Chronic Obstructive Pulmonary Disease (COPD) and Obesity Hypoventilation Syndrome (OHS) patients. By enhancing sleep comfort, adherence to ventilation will increase which, in turn, will improve ventilatory failure, quality of life and reduce length of admission during initiation of therapy. We aim to incorporate this technology into routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over the age of 16 years.
2. Patients with confirmed diagnosis of Duchenne Muscular dystrophy or Chronic Obstructive Pulmonary Disease or Obesity Hypoventilation Syndrome.
3. Patients with evidence of nocturnal hypoventilation with an arterial carbon dioxide partial pressure of >6.0 kPa in the morning.
4. Patients with evidence of hypercapnic respiratory failure with an arterial carbon dioxide partial pressure of >6.0 kPa during the day.
5. No prior domiciliary ventilation.

Exclusion Criteria:

1. Patients with other co-morbidities e.g. cancer or cardiac failure.
2. Patients with muscular weakness but an unconfirmed diagnosis of Duchenne Muscular Dystrophy, Obesity Hypoventilation Syndrome or Chronic Obstructive Pulmonary Disease.
3. Patients who have had an acute illness within the last 4 weeks prior to starting assessment for ventilation.
4. Patients who have an abnormal bleeding tendency (INR or APTTr >1.4 or platelets <100).
5. Patients with a psychological, social or geographical situation that would impair compliance with the project.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-01; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Adherence with ventilation | 3 months
  Data on patient reported compliance and ventilator recorded compliance will be collected.

SECONDARY OUTCOMES:
health related quality of life | 3 month
  SRI, RAND-36, visual analogue scores, St. George's respiratory questionnaire
length of hospital stay for initiation of home mechanical ventilation | 3 months
gas exchange | 3 months
  overnight oximetry, overnight capnography,arterial oxygenation, arterial carbon dioxide

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Guy's and St. Thomas' NHS Trust, London
  - Royal Brompton Hospital, London